CLINICAL TRIAL: NCT00383084
Title: Lifestyle Physical Activity for Fibromyalgia
Brief Title: Lifestyle Physical Activity to Reduce Pain and Fatigue in Adults With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01AR053168 (NIH); R01AR053168 (NIH); AR053168-01-A1
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2013-07-01 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Fibromyalgia
Keywords: Pain; Physical Activity; Fatigue; Lifestyle Activity
MeSH Terms: conditions — Fibromyalgia; Pain; Motor Activity; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Group 1 participants will take part in 30 minutes total of self-selected lifestyle physical activity throughout the day, 5 to 7 days per week. Twice a month, they will attend group sessions designed to help participants develop and maintain a more physically active lifestyle. Goal setting, self-monitoring, and pain management will be discussed at these sessions.
  Interventions: Behavioral: Lifestyle physical activity (LPA)
- 2 (Active Comparator): Group 2 participants will attend monthly fibromyalgia educational sessions, which will focus on understanding the symptoms of FM, learning to manage pain and fatigue, and developing self-help strategies.
  Interventions: Behavioral: Fibromyalgia education

INTERVENTIONS:
Behavioral: Lifestyle physical activity (LPA) — Bi-weekly, 60-minute group sessions spread over 12 weeks. Participants will receive education on how to increase their daily physical activity, goal setting, problem solving strategies to overcome barriers to being more physically active, and finding new ways to integrate short bouts of LPA into their daily lives.
  Arms: 1
Behavioral: Fibromyalgia education — Participants will meet monthly for 1.5 to 2 hours for a total of 3 months. The sessions will be divided into three components: (1) education, (2) question and answer, and (3) social support.
  Arms: 2

SUMMARY:
The purpose of this study is to determine the effect of 3 months of daily, 30-minute lifestyle physical activity on pain and fatigue in inactive adults with fibromyalgia (FM).

DETAILED DESCRIPTION:
FM is characterized by muscle pain, fatigue, and "tender points," specific places on the body that hurt when pressure is applied. Individuals with FM may also experience trouble sleeping, morning stiffness, headaches, and mood disorders. The exact cause of FM is unknown, and currently, there is no cure. While exercise improves the symptoms of FM, pain and fatigue often prevent individuals from beginning an exercise regimen in the first place. Because of the known benefits of exercise on FM, it is important to find new ways for individuals with FM to increase their physical activity. Lifestyle physical activity, which involves any type of moderate-intensity activity such as walking, housecleaning, shopping, and gardening, may be more doable than structured exercise for individuals with FM. Also, lifestyle physical activity accumulated in short bouts over time can be as effective as single exercise sessions in producing health benefits. The purpose of this study is to determine the effect of daily 30-minute lifestyle physical activity performed throughout the day on pain and fatigue in sedentary adults with FM.

This study will last 12 weeks. Participants will be randomly assigned to one of two groups. Group 1 participants will take part in 30 minutes total of self-selected lifestyle physical activity throughout the day, 5 to 7 days per week. Twice a month, they will attend group sessions designed to help participants develop and maintain a more physically active lifestyle. Goal setting, self-monitoring, and pain management will be discussed at these sessions. Group 2 participants will attend monthly FM educational sessions, which will focus on understanding the symptoms of FM, learning to manage pain and fatigue, and developing self-help strategies.

Throughout the study, both Group 1 and 2 participants will wear a wristwatch-sized device that will track their physical activity and record pain and fatigue levels. Evaluations will occur at baseline, Week 12, and 6 and 12 months after Week 12 for all participants. At each of these time points, participants will complete questionnaires, and undergo pain evaluations, fitness testing, and a tender point examination.

ELIGIBILITY:
Inclusion Criteria:

* Meets American College of Rheumatology (ACR) criteria for FM
* Inactive at study entry
* Willing to become more physically active
* Understands and willing to follow study recommendations regarding lifestyle modification
* Able to participate in the study for 2 years
* Agrees to not make any changes to current FM-related treatments

Exclusion Criteria:

* Any comorbidity that may worsen a participant's physical functioning, independent of FM (e.g., significant cardiovascular disease, history of arrhythmias, morbid obesity, autoimmune diseases, uncontrolled or untreated hypertension, significant renal or prostate disease, stroke, seizure disorder, any other significant neurological diseases)
* Significant peripheral neuropathy
* Any current psychiatric disorder that involves a history of psychosis, including schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, bipolar disorder, or severe personality disorder. Participants with mood disorder are not excluded.
* Alcohol or substance abuse within the 2 years prior to study entry
* Current suicide risk or suicide attempt within the 2 years prior to study entry
* Severe physical disability that may interfere with physical activity
* Currently participates in structured exercise or plans to participate in an exercise program
* Any investigational medications or devices within 4 weeks prior to study entry
* Any expected life change, such as relocation, within the next 2 years that may prevent study participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2006-09 (Actual); Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Fontaine, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Culos-Reed SN, Brawley LR. Fibromyalgia, physical activity, and daily functioning: the importance of efficacy and health-related quality of life. Arthritis Care Res. 2000 Dec;13(6):343-51. doi: 10.1002/1529-0131(200012)13:63.0.co;2-p. PMID 14635309
- [Background] Karper WB, Jannes CR, Hampton JL. Fibromyalgia syndrome: the beneficial effects of exercise. Rehabil Nurs. 2006 Sep-Oct;31(5):193-8. doi: 10.1002/j.2048-7940.2006.tb00135.x. PMID 16948441
- [Background] Oliver K, Cronan TA. Correlates of physical activity among women with fibromyalgia syndrome. Ann Behav Med. 2005 Feb;29(1):44-53. doi: 10.1207/s15324796abm2901_7. PMID 15677300
- [Derived] Campbell CM, McCauley L, Bounds SC, Mathur VA, Conn L, Simango M, Edwards RR, Fontaine KR. Changes in pain catastrophizing predict later changes in fibromyalgia clinical and experimental pain report: cross-lagged panel analyses of dispositional and situational catastrophizing. Arthritis Res Ther. 2012 Oct 25;14(5):R231. doi: 10.1186/ar4073. PMID 23098173
- [Derived] Fontaine KR, Conn L, Clauw DJ. Effects of lifestyle physical activity in adults with fibromyalgia: results at follow-up. J Clin Rheumatol. 2011 Mar;17(2):64-8. doi: 10.1097/RHU.0b013e31820e7ea7. PMID 21325963
- [Derived] Fontaine KR, Conn L, Clauw DJ. Effects of lifestyle physical activity on perceived symptoms and physical function in adults with fibromyalgia: results of a randomized trial. Arthritis Res Ther. 2010;12(2):R55. doi: 10.1186/ar2967. Epub 2010 Mar 30. PMID 20353551

RESULTS

PARTICIPANT FLOW:
Groups:
- Lifestyle Physical Activity: Group 1 participants will take part in 30 minutes total of self-selected lifestyle physical activity throughout the day, 5 to 7 days per week. Twice a month, they will attend group sessions designed to help participants develop and maintain a more physically active lifestyle. Goal setting, self-monitoring, and pain management will be discussed at these sessions.
- Education: Group 2 participants will attend monthly fibromyalgia educational sessions, which will focus on understanding the symptoms of FM, learning to manage pain and fatigue, and developing self-help strategies.
Period: Overall Study
Arm/Group | Lifestyle Physical Activity | Education
Started | 46 | 38
Completed | 34 | 28
Not Completed | 12 | 10
Not completed — Withdrawal by Subject | 12 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lifestyle Physical Activity | Education | Total
Number analyzed (Participants) | 46 | 38 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 38 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (11.6) | 49 (10.2) | 47.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 38 | 81
  Male | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 46 | 38 | 84

OUTCOME MEASURES:

1. Primary Outcome: Ambulatory Pain (Higher Values Indicate Greater Pain)
Description: 0 to 100 pain rating, higher numbers indicate greater pain
Time Frame: Baseline and after 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Physical Activity | Education
Number analyzed (Participants) | 46 | 38
units on a scale
  Baseline | 54.6 (25.6) | 58.9 (25)
  After 12 Weeks | 46.3 (24.2) | 62.4 (24.5)

2. Primary Outcome: Ambulatory Fatigue, Higher Values Indicate Greater Fatigue
Description: 0-100 fatigue ratings, higher scores indicative of greater levels of fatigue
Time Frame: Baseline and after 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Physical Activity | Education
Number analyzed (Participants) | 46 | 38
units on a scale
  Baseline | 51.9 (9.3) | 52.3 (9.1)
  After 12 Weeks | 50.6 (9.9) | 51.4 (10.1)

3. Secondary Outcome: Number of Tender Points on the Body
Description: Number of tender points on physical examination (maximum number is 18)
Time Frame: Baseline and after 12-weeks
Measure: Mean (Standard Deviation); unit: tender points
Arm/Group | Lifestyle Physical Activity | Education
Number analyzed (Participants) | 46 | 38
tender points
  Baseline | 16.2 (2.3) | 16.1 (3.2)
  After 12 Weeks | 16 (2.3) | 16.8 (2.0)

4. Secondary Outcome: Functional Capacity (Higher Scores Indicative of Poorer Functioning)
Description: Fibromyalgia Impact Questionnaire (a higher total score indicates poorer functioning). The range of possible scores is 0 to 100
Time Frame: Baseline and after 12-weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle Physical Activity | Education
Number analyzed (Participants) | 46 | 38
units on a scale
  Baseline | 67.5 (12) | 69.7 (13.4)
  After 12 Weeks | 56.7 (20.6) | 67 (18.6)

ADVERSE EVENTS:
Arm/Group | Lifestyle Physical Activity | Education
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/38
Other Adverse Events (participants affected / at risk) | 0/46 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Restriction type: embargo of 60 days or less